CLINICAL TRIAL: NCT06982976
Title: Efficacy and Safety of Photodynamic Therapy for Cervical and Vaginal Intraepithelial Neoplasia:A Multicenter Prospective Cohort Study
Brief Title: Efficacy and Safety of Photodynamic Therapy for Cervical and Vaginal Intraepithelial Neoplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-M2023505; 2022YFB3604704 (Other Grant/Funding Number: Ministry of Science and Technology of the People's Republic of China)
Record Dates: First submitted 2025-04-29; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Precancerous Cervical Lesion
Keywords: ALA-PDT; HPV; CIN; VAIN

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALA-PDT (Other): Patients choose PDT to treat the disease
  Interventions: Procedure: ALA-PDT

INTERVENTIONS:
Procedure: ALA-PDT — use ALA_PDT to treat the disease

SUMMARY:
To investigate the efficacy and safety of photodynamic therapy (20% 5-amino-ketovalerate 630nm red light) in the treatment of cervical and vaginal intraepithelial neoplasia in women in the real world.

ELIGIBILITY:
Inclusion Criteria:

* cervical/vaginal high-grade squamous intraepithelial lesions (HSILs) confirmed by colposcopy and pathological biopsy (CIN2 /CIN3 and/or VaIN2/ VaIN3) or persistent CIN1/VaIN1 lasting for more than one year with a strong willingness to treat;
* colposcopy was adequate, and analysable colposcopy images were retained;
* endocervical curettage (ECC) did not suggest higher-grade lesions.

Exclusion Criteria:

* coexistence or suspicion of cancer;
* porphyria or suspected allergies to red and blue light;
* severe medical comorbidities；

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the treatment | 1 month after the treatment
  colposcopy and biopsy will be performed one month after the treatment. Patients will be categorised as having complete remission(CR) if biopsy confirmed LSIL. If CIN 2/VAIN 2 was found after the first course of PDT, it would be categorised as partial remission(PR) if they are CIN3/VAIN3 before treatment. Those with the same grade were categorised as persistent disease(PD).
  The proportion of CR and PR after PDT treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Unniversity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT06982976/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT06982976/ICF_001.pdf